CLINICAL TRIAL: NCT05727371
Title: Multicenter, Randomized Double-blind Study to Compare the Safety and Performance of a Combination of A-PRP and XLHA Prepared With the RegenMatrix Medical Device, to Hylan G-F 20 XLHA and Placebo to Treat Moderate/Severe Knee Osteoarthritis
Brief Title: Combination of PRP and XLHA Prepared With RegenMatrix Medical Device To Treat Moderate to Severe Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RegenLab France SAS (Industry)
Responsible Party: Sponsor
Organization: Regen Lab SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-A01514-39
Record Dates: First submitted 2023-01-09; First posted 2023-02-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
Keywords: platelet-rich plasma; cross-linked hyaluronic acid; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RegenMatrix-PRP-XLHA (Experimental): Patients randomized in this group will receive a single injection of a combination of platelet-rich plasma plus cross-linked hyaluronic acid, prepared with the medical device RegenMatrix.
  Interventions: Combination Product: Regen Matrix-PRP-XLHA
- Hylan G-F 20 (Active Comparator): Patients randomized in this group will receive a single injection of cross-linked hyaluronic acid Hylan G-F 20 (Synvisc-One®).
  Interventions: Device: Hylan G-F 20
- Placebo (Placebo Comparator): Patients randomized in this group will receive a single injection of saline solution (0.9% NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: Regen Matrix-PRP-XLHA — Single intra-articular injection at Day 0
  Arms: RegenMatrix-PRP-XLHA
Device: Hylan G-F 20 — Single intra-articular injection at Day 0
  Arms: Hylan G-F 20
Drug: Placebo — Single intra-articular injection at Day 0
  Arms: Placebo

SUMMARY:
In this clinical trial the investigator assess the safety and efficacy of a single injection of a combination of cross-linked hyaluronic acid (HA) with autologous platelet-rich plasma (PRP) obtained with the RegenMatrix medical device to improve symptoms of moderate to severe knee osteoarthitis (grade III-IV Kellgren-Lawrence).

DETAILED DESCRIPTION:
In this multicenter, randomized, double-blind, three-arm study, the investigator propose to evaluate the safety and efficacy at Day0, Month1, Month3 and Month6 of a single intra-articular injection of a combination RM-PRP-XLHA (experimental treatment: combination of cross-linked HA and PRP obtained with the RegenMatrix medical device) against Hylan G-F 20 (reference treatment) and placebo for the treatment of moderate to severe knee osteoarthritis.

The symptomatic benefit will be evaluated in terms of pain reduction and improvement of patient's quality of life. The functional benefit of the treatment will also be evaluated, on a reduced number of participants, by a gait analysis, performed only in the coordinating centre.

The medical device RegenMatrix is an adaptation of the medical device Cellular Matrix (certified since 2013,CE2797). It differs from the latter only for by presence of cross-linked HA instead of linear HA, and is therefore particularly suitable for the treatment of moderate to severe knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Tibiofemoral knee osteoarthrosis according to ACR criteria
* Tibiofemoral knee osteoarthrosis grade 3-4 according to the Kellgren & Lawrence grading scale, as defined on knee radiographs (less than 3 months old: face view, schuss view, profile and patellar axial view at 30°)
* Symptomatic knee osteoarthrosis as evidenced by pain on walking (WOMAC A1 assessed in the last 24 hours on a scale of 0 to 100 mm: 50 ≤ DM 90 or reduced joint function (WOMAC C total score assessed or within the previous 24 hours based on a scale of 0-100-mm: 50 ≤ WOMAC C ≤ 90)
* Patient able to understand the requirements of the trial and who has signed a free and informed consent prior to study entry
* Patient able to read and understand the written instructions
* Patient able to complete the self-assessment questionnaires

Exclusion Criteria:

* Tibiofemoral knee osteoarthrosis grade I or II according to the Kellgren and Lawrence grading scale
* Knee surgery planned in the next 6 months
* Patient affected by autoimmune disease (rheumatoid arthritis, lupus, Hashimoto's disease and Bechterew's syndrome)
* Chronic inflammatory rheumatism other than arthritis (polyarthrosis, etc.)
* Patient affected by a knee infection in the past 6 months
* Clinical signs of local knee inflammation (redness or warmth of the knee joint)
* Last PRP or PRP/HA injection received in the last year
* Last viscosupplementation received in the past 6 months
* Last corticosteroid injection received in the past 3 months
* Use of gluco-corticosteroids (except inhaled) and level III analgesics in the last 3 months and non-steroidal anti-inflammatory drug in the last 2 weeks
* Treatment with AAAL initiated within the last 6 months
* History of allergy to hyaluronic acid
* Hematologic or clotting disorders (thrombocytopenia) or blood coagulation (deficit-blood dyscrasia)
* Patients with coagulation times outside the reference values
* Anemia (HGB<10 g/dl)
* Venous or lymphatic stasis in the corresponding limb
* Malignant diseases (especially bone or haematological)
* Patients with serious, no-stabilized pathologies (cardiovascular disease, active peptic ulcer, digestive hemorrhage)
* Acute infection
* Patients with cancer or with an immuno-deprassant treatment ongoing
* Participation in another clinical trial for osteoarthritis of the knee in the last year
* Participation in another clinical trial, ongoing or completed within the last 3 months
* Patient unable to comply with the constraints of the protocol, in particular a patient whose mental state does not allow him/her to patient's mental state does not allow him/her to understand the nature, objectives and possible consequences of the study
* Pregnant or breastfeeding women or women who expect to become pregnant during the study
* Any other reason which may interfere with the proper conduct of the study, in the investigator's opinion

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Variation in the osteoarthritis related pain | 6 months (Day 0 - Month 6)
  It will be assessed by the mean difference in the WOMAC A score on a 100-mm VAS overtime

SECONDARY OUTCOMES:
Variation in the overall osteoarthritis related pain | M1 and M3 (Day 0-Month 1; Day 0 - Month 3)
  It will be assessed by the mean difference in the WOMAC A score on a 100-mm VAS overtime
Variation of joint stiffness after the first awakening and later in the day | Month 1, Month 3 and Month 6 (Day 0-Month 1; Day 0-Month 3; Day 0-Month 6)
  It will be assessed by the mean difference in the WOMAC B score overtime
Variation of joint function during daily activity | Month 1, Month 3 and Month 6 (Day 0-Month 1; Day 0-Month 3; Day 0-Month 6)
  It will be assessed by the mean difference in the WOMAC C score overtime
Variation in the osteoarthritis related symptoms | Month 1, Month 3 and Month 6 (Day 0-Month 1; Day 0-Month 3; Day 0-Month 6)
  It will be assessed by the mean difference in the total WOMAC score Month 1, Month 3 and M6 (D0-M1; D0-M3; D0-M6)
Variation of patient's quality of life | Month 1, Month 3 and Month 6 (Day 0-Month 1; Day 0-Month 3; Day 0-Month 6)
  It will be assessed by the SF-12 questionnaire
Pain, function, patient's general assessment | Month 1, Month 3 and Month 6 (Day 0-Month 1; Day 0-Month 3; Day 0-Month 6)
  It will be assessed by the% of OMERACT-OARSI responders
Assessment of the minimal meaningful change according to the patient's perception | Month 1, Month 3 and Month 6 (Day 0-Month 1; Day 0-Month 3; Day 0-Month 6)
  The Minimal Clinically Important Improvement (MCII) will be assessed on the basis of the answers to the WOMAC questionnaire.
Assessment of the highest level of symptom beyond which patients consider themselves well. | Month 1, Month 3 and Month 6 (D0-Month 1; Day 0-Month 3; Day 0-Month 6)
  The Patient Acceptable Symptom State (PASS) will be assessed on the basis of the answers to the WOMAC questionnaire.
Rescue medication | Month 1, Month 3 and Month 6 (Day 0-Month 1; Day 0-Month 3; Day 0-Month 6)
  Consumption of level 1 and 2 painkillers, NSAIDs and corticosteroids

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ornetti, MD, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (13):
- France (13):
  - Hopital Le Bocage Chru, Dijon, DE
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - CHU Henri Mondor APHP, Créteil
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - CHU Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Hopital Lapeyronie, Montpellier
  - CHU Nantes Hôtel - Dieu, Nantes
  - Ch de Narbonne, Narbonne
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Antoine, Paris
  - Hopital Maison Blanche, Reims
  - Clinique Medipole Garonne, Radiologie Interventionnelle 45 Rue Gironis, Toulouse

IPD SHARING:
Plan to Share IPD: No